CLINICAL TRIAL: NCT02593305
Title: Dietary Nitrate Supplementation and Physiological Function in Older Adults
Brief Title: Dietary Nitrate and Physiological Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Darren P Casey (Other)
Collaborators: Neogenis Laboratories (Other)
Responsible Party: Sponsor-Investigator, Darren P Casey, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 201507735
Record Dates: First submitted 2015-10-27; First posted 2015-11-02 (Estimated); Results first posted 2019-10-14 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-09

CONDITIONS: Aging
Keywords: nitrate; blood flow; blood pressure; vascular function; hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Beetroot crystals (nitrate), then placebo (Experimental): Participants will receive a nitrate rich beetroot powder (10g/day) for 4 weeks. After a washout period of 4 weeks, they will then receive the placebo (beetroot powder, no nitrate) for 4 weeks.
  Interventions: Dietary Supplement: Super Beets; Dietary Supplement: Super Beets Placebo
- Placebo, then beetroot crystals (nitrate) (Experimental): Participants will receive a beetroot powder placebo (no nitrate) for 4 weeks. After a 4 week washout period, they will receive the nitrate rich beetroot powder for 4 weeks.
  Interventions: Dietary Supplement: Super Beets; Dietary Supplement: Super Beets Placebo
- Young Comparison (No Intervention): Young control group, used for age-related comparisons. This group did not go through any intervention.

INTERVENTIONS:
Dietary Supplement: Super Beets — Nitrate rich beetroot powder (10g/day) for 4 weeks
  Other Names: Beetroot crystals
  Arms: Beetroot crystals (nitrate), then placebo; Placebo, then beetroot crystals (nitrate)
Dietary Supplement: Super Beets Placebo — Nitrate deficient beetroot powder (10g/day) for 4 weeks
  Other Names: Beetroot crystals no nitrate
  Arms: Beetroot crystals (nitrate), then placebo; Placebo, then beetroot crystals (nitrate)

SUMMARY:
The main purpose/s of this study is to examine the effects of 4 weeks of dietary nitrate supplementation on peripheral chemoreceptor sensitivity, spontaneous baroreflex sensitivity, and blood pressure responsiveness to a variety of physiological stressors in older healthy adults. We will also examine the effect of dietary nitrate supplementation on measures of central artery stiffness and aortic blood pressure in older adults. Lastly, we will also recruit a group of young subjects in order to help characterize the age-related changes associated with the physiological outcome measures of the present study.

DETAILED DESCRIPTION:
1 in 3 adults in the U.S. have hypertension which is known to increase the risk of heart disease and stroke. Blood pressure regulation is mediated by many factors including but not limited to metabolic factors, pressure/stretch sensing receptors located in the aorta and carotid arteries, endothelial cell function, and kidney function (via water and sodium absorption/excretion). It has been shown that many of these regulatory mechanisms are altered and/or become dysfunctional with aging. Specifically older adults commonly demonstrate a decreased sensitivity in pressure receptors and/or endothelial dysfunction. Additionally with aging, there is an increase in sympathetic nervous system activity and arterial stiffness which can contribute to higher blood pressure. The important vasodilator, nitric oxide (NO), has been implicated as a key signaling molecule involved in several of the mechanisms in blood pressure regulation outlined above. A decreased NO production or bioavailability is thought to contribute to several of the physiologic changes that come with aging. Therefore, the overall aim of this study is to use a randomized, double-blind crossover, placebo controlled study to examine the effects of acute dietary nitrate supplementation (to boost bioavailable NO) on various parameters of blood pressure regulation and responsiveness in normal healthy older adults. Our main hypothesis is that 4 weeks of dietary nitrate supplementation will decrease the blood pressure responses in older adults in response to a variety of physiological stressors.

ELIGIBILITY:
Two separate age groups were included.

Inclusion Criteria:

* Healthy young adults 18-35 years of age (comparison group)
* Healthy older adults 60-85 years of age (intervention group)

Exclusion Criteria:

* Hypertension, hyperlipidemia, current smoker or smoker within the last year, heart disease, diabetes, Chronic obstructive pulmonary disease, asthma, sleep apnea, Raynaud's disease, body mass index (BMI) > 30 kg/m2, allergy medication, clinical depression, autonomic disorders and other conditions or medications that might normally alter cardiovascular function, exercise tolerance, and/or blood pressure responses.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-10; Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darren Casey, PhD., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nitrate First Arm: Subjects consumed beet root juice with nitrate for 4 weeks during the first arm of the study. After a 4 week washout period, subjects consumed beetroot juice without nitrate (placebo) for 4 weeks.
- Placebo First Arm: Subjects consumed beet root juice without nitrate (placebo) for 4 weeks during the first arm of the study. After a 4 week washout period, subjects consumed beetroot juice with nitrate for 4 weeks.
- Young Comparison Group: Young subjects only completed a single experimental visit and no intervention. Data from young were used for age-related comparisons at baseline.
Period: Baseline 1
Arm/Group | Nitrate First Arm | Placebo First Arm | Young Comparison Group
Started | 7 | 6 | 10
Completed | 7 | 6 | 10
Not Completed | 0 | 0 | 0
Period: Post 1
Arm/Group | Nitrate First Arm | Placebo First Arm | Young Comparison Group
Started | 7 | 6 | 10
Completed | 7 | 6 | 0
Not Completed | 0 | 0 | 10
Not completed — Comparison only group. No intervention. | 0 | 0 | 10
Period: Baseline 2
Arm/Group | Nitrate First Arm | Placebo First Arm | Young Comparison Group
Started | 7 | 6 | 0
Completed | 7 | 6 | 0
Not Completed | 0 | 0 | 0
Period: Post 2
Arm/Group | Nitrate First Arm | Placebo First Arm | Young Comparison Group
Started | 7 | 6 | 0
Completed | 7 | 6 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Young Comparison Group: Young control group, used for age-related comparisons. This group did not go through any intervention.
- Total: Total of all reporting groups
Arm/Group | Nitrate First Arm | Placebo First Arm | Young Comparison Group | Total
Number analyzed (Participants) | 7 | 6 | 10 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 10 | 11
  >=65 years | 6 | 6 | 0 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Row population reflect each distinct age group. Row older adults =13 subjects. Row young adults = 10 subjects. Together the two age groups (rows) total the overall 23 subjects enrolled in the study.
  years
    Older Adults: number analyzed (Participants) | 7 | 6 | 0 | 13
    Older Adults | 68 (3) | 66 (2) |  | 67 (3)
    Young Adults: number analyzed (Participants) | 0 | 0 | 10 | 10
    Young Adults |  |  | 25 (4) | 25 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 5 | 11
  Male | 5 | 2 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 6 | 10 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 6 | 9 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 10 | 23
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Row population reflect each distinct age group. Row older adults =13 subjects. Row young adults = 10 subjects. Together the two age groups (rows) total the overall 23 subjects enrolled in the study.
  kg/m^2
    Older Adults: number analyzed (Participants) | 7 | 6 | 0 | 13
    Older Adults | 26 (4) | 25 (3) |  | 26 (3)
    Young Adults: number analyzed (Participants) | 0 | 0 | 10 | 10
    Young Adults |  |  | 24 (3) | 24 (3)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: Row population reflect each distinct age group. Row older adults =13 subjects. Row young adults = 10 subjects. Together the two age groups (rows) total the overall 23 subjects enrolled in the study.
  mmHg
    Older Adults: number analyzed (Participants) | 7 | 6 | 0 | 13
    Older Adults | 126 (12) | 118 (5) |  | 122 (10)
    Young Adults: number analyzed (Participants) | 0 | 0 | 10 | 10
    Young Adults |  |  | 119 (8) | 119 (8)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: Row population reflect each distinct age group. Row older adults =13 subjects. Row young adults = 10 subjects. Together the two age groups (rows) total the overall 23 subjects enrolled in the study.
  mmHg
    Older Adults: number analyzed (Participants) | 7 | 6 | 0 | 13
    Older Adults | 76 (5) | 75 (6) |  | 76 (5)
    Young Adults: number analyzed (Participants) | 0 | 0 | 10 | 10
    Young Adults |  |  | 72 (5) | 72 (5)
Glucose [Mean (Standard Deviation); unit: mg/dl] — Population: Row population reflect each distinct age group. Row older adults =13 subjects. Row young adults = 10 subjects. Together the two age groups (rows) total the overall 23 subjects enrolled in the study.
  mg/dl
    Older Adults: number analyzed (Participants) | 7 | 6 | 0 | 13
    Older Adults | 97 (7) | 96 (4) |  | 96 (5)
    Young Adults: number analyzed (Participants) | 0 | 0 | 10 | 10
    Young Adults |  |  | 89 (5) | 89 (5)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dl] — Population: Row population reflect each distinct age group. Row older adults =13 subjects. Row young adults = 10 subjects. Together the two age groups (rows) total the overall 23 subjects enrolled in the study.
  mg/dl
    Older Adults: number analyzed (Participants) | 7 | 6 | 0 | 13
    Older Adults | 171 (40) | 184 (31) |  | 177 (35)
    Young Adults: number analyzed (Participants) | 0 | 0 | 10 | 10
    Young Adults |  |  | 153 (22) | 153 (22)
HDL [Mean (Standard Deviation); unit: mg/dl] — Population: Row population reflect each distinct age group. Row older adults =13 subjects. Row young adults = 10 subjects. Together the two age groups (rows) total the overall 23 subjects enrolled in the study.
  mg/dl
    Older Adults: number analyzed (Participants) | 7 | 6 | 0 | 13
    Older Adults | 57 (19) | 49 (21) |  | 53 (19)
    Young Adults: number analyzed (Participants) | 0 | 0 | 10 | 10
    Young Adults |  |  | 60 (15) | 60 (15)
LDL [Mean (Standard Deviation); unit: mg/dl] — Population: Row population reflect each distinct age group. Row older adults =13 subjects. Row young adults = 10 subjects. Together the two age groups (rows) total the overall 23 subjects enrolled in the study.
  mg/dl
    Older Adults: number analyzed (Participants) | 7 | 6 | 0 | 13
    Older Adults | 98 (33) | 107 (33) |  | 102 (32)
    Young Adults: number analyzed (Participants) | 0 | 0 | 10 | 10
    Young Adults |  |  | 82 (23) | 82 (23)
Triglycerides [Mean (Standard Deviation); unit: mg/dl] — Population: Row population reflect each distinct age group. Row older adults =13 subjects. Row young adults = 10 subjects. Together the two age groups (rows) total the overall 23 subjects enrolled in the study.
  mg/dl
    Older Adults: number analyzed (Participants) | 7 | 6 | 0 | 13
    Older Adults | 84 (39) | 144 (84) |  | 111 (69)
    Young Adults: number analyzed (Participants) | 0 | 0 | 10 | 10
    Young Adults |  |  | 53 (12) | 53 (12)

OUTCOME MEASURES:

1. Primary Outcome: Change in Carotid Chemosensitivity Following 4 Weeks of Dietary Nitrate Supplementation and Placebo in Older Adults
Description: Carotid chemosensitivity examined by measuring hypoxia ventilatory responsiveness in older adults before and after 4 weeks of beet root juice supplementation and placebo. Chemoreflex sensitivity was quantified as the change in ventilation in relation to the change in pulse oxygen saturation.
Time Frame: Pre and post 4 weeks dietary nitrate supplementation and pre and post 4 weeks of placebo.
Measure: Mean (Standard Error); unit: L/min/%SpO2
Groups:
- Nitrate Pre: Subjects randomized to the nitrate group for 4 weeks. Values reflect pre intervention measures.
- Nitrate Post: Subjects randomized to the nitrate group for 4 weeks. Values reflect post intervention measures.
- Placebo Pre: Subjects randomized to the placebo group for 4 weeks. Values reflect pre intervention measures.
- Placebo Post: Subjects randomized to the placebo group for 4 weeks. Values reflect post intervention measures.
Arm/Group | Nitrate Pre | Nitrate Post | Placebo Pre | Placebo Post
Number analyzed (Participants) | 13 | 13 | 13 | 13
L/min/%SpO2 | -0.13 (0.04) | -0.05 (0.02) | -0.10 (0.05) | -0.11 (0.05)

2. Primary Outcome: Change in Systolic Blood Pressure During Metaboreflex Testing Following 4 Weeks of Dietary Nitrate Supplementation and Placebo in Older Adults.
Description: Muscle metaboreflex examined by measuring systolic blood pressure responses to ischemic isometric muscle contraction in older adults before and after 4 weeks of beet root juice supplementation and placebo.
Time Frame: Pre and post 4 weeks dietary nitrate supplementation and pre and post 4 weeks of placebo.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Nitrate Pre | Nitrate Post | Placebo Pre | Placebo Post
Number analyzed (Participants) | 13 | 13 | 13 | 13
mmHg | 19.2 (2.1) | 13 (2.5) | 16.1 (1.8) | 17 (1.9)

ADVERSE EVENTS:
Time Frame: The length of study enrollment of each older subject (~3 months). Young subjects only completed one single study visit.
Groups:
- Nitrate: Subjects consumed beet root juice with nitrate for 4 weeks.
- Placebo: Subjects consumed beet root juice without nitrate (placebo) for 4 weeks.
- Young Comparison Group: Subjects completed one single study visit.
Arm/Group | Nitrate | Placebo | Young Comparison Group
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/10
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/10

LIMITATIONS AND CAVEATS:
All subjects (young and older) completed the initial study visit. The young adults were used as a comparison group only and did not go through any intervention. The older adults underwent the intervention and completed a total of four study visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2016-07-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT02593305/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2015-07-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT02593305/Prot_SAP_001.pdf